CLINICAL TRIAL: NCT01644851
Title: Cognitive Training for PTSD: Effects on Cognitive, Emotional, and Brain Function
Brief Title: Cognitive Training for Post Traumatic Stress Disorder: Effects on Cognitive, Emotional, and Brain Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Principal Investigator, Robin Aupperle, Assistant Professor, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMKC SS11-212e
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Posttraumatic Stress Disorders
Keywords: veterans; neuropsychology; neuroimaging; attention; working memory; inhibition; magnetic resonance imaging, functional; trauma; stress; anxiety; emotion; prefrontal cortex
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Inhibition, Psychological; Wounds and Injuries; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Executive function training (Experimental): Executive function training
  Interventions: Behavioral: Executive function training
- Word game training (Placebo Comparator): Computer-based training in tasks related to verbal processing.

INTERVENTIONS:
Behavioral: Executive function training — Computer-based training in executive functions, administered via www.lumosity.com website.
  Arms: Executive function training

SUMMARY:
The purpose of this pilot study is to determine the effects of computer-based training in executive functioning compared to word games on cognitive and emotional aspects of combat-related PTSD.

DETAILED DESCRIPTION:
Many posttraumatic stress disorder (PTSD) patients either choose not to complete or do not achieve optimal response to current first-line behavioral and pharmacologic treatments. Neurocognitive research points to the potential of novel treatments targeting dorsal prefrontal function and inhibition, attention, and working memory processes. This study investigates effects of computer-based training in executive functions compared to word games on cognitive and emotional aspects of combat-related PTSD. Paper-and-pencil questionnaires, interviews, computer-administered testing, and magnetic resonance imaging will be complete before and after the intervention. Results from this pilot study will provide information concerning feasibility and treatment potential of cognitive training for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* combat veterans who served in Operation Iraqi Freedom, Operation Enduring Freedom, or Operation New Dawn

Exclusion Criteria:

* enrolled in other active treatment protocols
* current substance abuse or dependence
* current suicidal ideation
* diagnosis of a neurological disorder
* history of moderate to severe traumatic brain injury

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Neural activity in prefrontal regions during cognitive and emotional processing measured by functional magnetic resonance imaging. | change from baseline to after 6 weeks of training

SECONDARY OUTCOMES:
Cognitive functioning as measured by neuropsychological assessment. | change from baseline to after 6 weeks of training

OTHER OUTCOMES:
Clinical PTSD symptoms as measured by the Clinician Administered PTSD Scale (CAPS). | change from baseline to after 6 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Robin Aupperle, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- Univesity of Missouri - Kansas City, Kansas City, Missouri, United States